CLINICAL TRIAL: NCT01271140
Title: High Dose Insulin Therapy to Improve Liver Function in Patients With HCV Liver Cirrhosis
Brief Title: High Dose Insulin Therapy to Improve Liver Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, peter metrakos, Director Multiorgan Transplant Program-MUHC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-086-BMA
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin/dextrose clamp (Experimental)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Intravenous insulin clamp at a rate of 2 mlu/kg/hr. In adition a titrating dose of 20% dextrose aiming to a blood glucose level of 4 - 5.5 mmol/l.
  Other Names: Hyperinsulinemic normoglycemic clamp

SUMMARY:
Insulin resistance is one of the key factors in defining a progressive course of chronic Hepatitis C virus (HCV) infection and hepatic fibrosis. Multiple trials have targeted insulin resistance as an adjuvant way to manage hepatitis C liver disease with promising results.

Long term therapy using high dose insulin was shown to significantly reduce insulin resistance in obese patients. In cardiac and critically ill patients, long term insulin was shown to produce better outcomes mainly by reducing the overt inflammatory response. Furthermore, initial results of ongoing trials are revealing more benefits of insulin therapy. Using the (hyperinsulinimic normoglycemic clamp) for eight hours on patients undergoing major liver resection was able to maximize their liver function post-operatively. This trial also demonstrated inhibition of the inflammatory response, improvement in liver glycogen, inhibition of apoptosis and stimulation of liver regeneration.

Putting in mind the potential ability of the liver to regenerate and regain better function. The anti-inflammatory properties of insulin therapy along with its ability to reduce insulin resistance over time has led us to see the potential benefits of using insulin therapy on patients with chronic hepatitis C virus liver cirrhosis. Insulin will target the pathophysiology of the disease at a cellular and a molecular level.

The investigators theorize that long-term high insulin therapy would be able to promote better liver function and slow down fibrosis and injury in this population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C positive adult patients (serum HCV antibody positive)
* MELD score 6-15 at the time of inclusion
* Viral genotype "non-3"
* Not on antiviral therapy

Exclusion Criteria:

* HBV or HIV co-infection
* Evidence of hepatocellular carcinoma at the start of the trial either by imaging and or AFP levels above 400
* Undetectable HCV viral load (using HCV PCR test)
* Recent infection or bleeding (in the last 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Liver status improvments (biochemical and histological) | 6 months

SECONDARY OUTCOMES:
Insulin resistance | 6 months
Inflammatory mediators | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Metrakos, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Helath Centre - (Royal Victoria Hospital), Montreal, Quebec, Canada